CLINICAL TRIAL: NCT01753999
Title: Obstructive Sleep Apnea in WTC Responders: Role of Nasal Pathology
Brief Title: Obstructive Sleep Apnea in World Trade Center Responders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: NYU Langone Health (Other)
Responsible Party: Principal Investigator, Jag Sunderram, MD, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012002164; 1U01OH010415-01 (NIH)
Record Dates: First submitted 2012-12-17; First posted 2012-12-21 (Estimated); Results first posted 2018-07-20 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: World Trade Center (WTC); nasal symptoms; nasal inflammation; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard CPAP (Active Comparator): Use of a standard CPAP (continuous positive airway pressure) device with constant pressure for 4 weeks to improve breathing during sleep
  Interventions: Device: Standard CPAP
- CPAP - Flex (Active Comparator): Use of CPAP-Flex (continuous positive airway pressure) device with decreased pressure during expiration for 4 weeks to improve breathing during sleep
  Interventions: Device: CPAP - Flex

INTERVENTIONS:
Device: Standard CPAP — Use of the REMstar Auto A-Flex in standard CPAP therapy mode
  Other Names: Philips Respironics REMstar Auto A-Flex
  Arms: Standard CPAP
Device: CPAP - Flex — Use of Philips Respironics REMstar Auto A-Flex in C-Flex mode
  Other Names: Philips Respironics REMstar Auto A-Flex
  Arms: CPAP - Flex

SUMMARY:
The goal of the study is to examine the possible underlying causes of sleep apnea (a disorder in which there are problems with breathing during sleep) in World Trade Center Responders. The study will look at the relationship between sleep apnea and various nose and throat conditions. Specifically, the study will look at upper airway disease (problems with the nose and throat), nasal inflammation, and nasal resistance (the amount of airflow through the nose). Subjects will have a physical exam and answer questions about nasal symptoms and sleeping problems. Nasal lavage (washing the inner nasal passages) will be performed on the subjects and markers of inflammation will be measured in the lavage fluid. Rhinomanometry (measuring the airflow through the nose) will also be performed to measure the degree of airflow obstruction. All subjects will be asked to perform in-home sleep apnea monitoring. Those subjects who are diagnosed with sleep apnea will test two treatment methods. Sleep apnea is treated by using a CPAP (continuous positive airway pressure) device. This device blows air into a mask worn by the patient during sleep. The two treatment methods that will be tested are the fixed pressure CPAP (pressure is constant during use) and CPAP-flex (pressure decreases when the subject exhales). Patients will be randomly assigned to one treatment method for one month then crossed to the other treatment method for the next month. The investigators will determine if patients with certain nasal conditions (high nasal resistance) are more likely to use CPAP-flex rather than CPAP.

DETAILED DESCRIPTION:
Following the World Trade Center (WTC) disaster, an estimated 40,000 individuals were exposed to significant amounts of dust while working in rescue, recovery and debris removal. A significant number of these responders have reported least one new or worsened upper airway respiratory symptom when examined in 2004 with 50% of responders continuing to have symptoms of chronic rhino-sinusitis or upper airway disease (UAD) in 2007. In addition, about 50% of those with UAD referred to our sleep center reported new onset snoring on their questionnaires immediately following their exposure and had unusually high prevalence of obstructive sleep apnea (OSA) that did not appear to be related to obesity, which is the usual risk factor for OSA. This suggests to us that mechanisms other than obesity may be important in the pathogenesis of OSA in these subjects. Given their chronic nasal symptoms they also provide a unique opportunity to examine the relationship between nasal pathology and OSA and test if nasal symptoms reported by the subjects in the WTC Health Program (WTCHP) are an indicator of increased nasal resistance due to nasal inflammation resulting from exposure to the WTC dust. Positive Airway Pressure (CPAP) is the standard therapy for OSA but despite its efficacy has poor adherence. Subjects with high nasal resistance (such as responders with UAD and OSA) may experience additional pressure during expiration at the upper airway resulting in greater difficulty in tolerating CPAP therapy than those who do not have high nasal resistance. Reduction of excess expiratory positive pressure by the modality known as Cflex™ during CPAP therapy (CPAPFlex) may improve comfort and adherence in these subjects without compromising CPAP efficacy. In the present proposal we will study responders enrolled at the Environmental and Occupational Health Sciences Institute of Robert Wood Johnson Medical School (RWJMS) and the NYU School of Medicine Clinical Center of Excellence at Bellevue Hospital

ELIGIBILITY:
Inclusion Criteria:

* Member of the World Trade Center Health Program at either the Environmental and Occupational Healthy Sciences Institute at Robert Wood Johnson Medical School in Piscataway, NJ, the New York University School of Medicine Clinical Center of Excellence at Bellevue Hospital in New York, NY, or the Icahn School of Medicine at Mount Sinai.

Exclusion Criteria:

* Gross skeletal alterations affecting the upper airway (nose and throat)
* Unstable chronic medical conditions known to affect Obstructive Sleep Apnea (congestive heart failure, stroke)
* Pregnancy or intent to become pregnant
* Habitual snoring or diagnosis of obstructive sleep apnea prior to 9/11/2001.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jag Sunderram, MD, Principal Investigator — Rutgers RWJMS; Indu Ayappa, PhD, Principal Investigator — NYUMC
Locations (3):
- United States (3):
  - Environmental and Occupational Health Sciences Institute, Piscataway, New Jersey
  - New York University School of Medicine Clinical Center of Excellence, New York, New York
  - Mount Sinai School of Medicine, New York, New York

REFERENCES:
- [Derived] Sunderram J, Ayappa I, Lu SE, Wang H, Black K, Twumasi A, Sanders H, Harrison D, Udasin I, Chitkara N, de la Hoz RE, Carson JL, Rapoport DM. PAP Adherence and Nasal Resistance. A Randomized Controlled Trial of CPAPflex versus CPAP in World Trade Center Responders. Ann Am Thorac Soc. 2021 Apr;18(4):668-677. doi: 10.1513/AnnalsATS.202009-1161OC. PMID 33202147
- [Derived] Ayappa I, Sunderram J, Black K, Twumasi A, Udasin I, Harrison D, Carson JL, Lu SE, Rapoport DM. A comparison of CPAP and CPAPFLEX in the treatment of obstructive sleep apnea in World Trade Center responders: study protocol for a randomized controlled trial. Trials. 2015 Sep 10;16:403. doi: 10.1186/s13063-015-0907-7. PMID 26357928

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between January 2013 and December 2016 at three World Trade Center Health Program Clinical Centers of Excellence (Rutgers University, Icahn School of Medicine at Mount Sinai, and New York University School of Medicine).
Pre-assignment Details: Subjects without OSA were excluded from the trial.
Groups:
- Standard CPAP Followed by CPAP-Flex: Participants were first treated with standard CPAP (continuous positive airway pressure with constant pressure) using a REMstar Auto A-flex in standard CPAP therapy mode for 4 weeks. The therapy mode was then switched to CPAP-Flex for 4 weeks. CPAP-Flex provides a decrease in pressure during expiration.
- CPAP-Flex Followed by Standard CPAP: Participants were treated with CPAP-Flex (continuous positive airway pressure with a decrease in pressure during expiration) using a REMstar Auto A-flex in C-Flex mode for 4 weeks. The therapy mode was then switched to standard CPAP for 4 weeks. Standard CPAP provides a constant pressure (no decrease after expiration).
Period: Period 1 - Initial Assignment
Arm/Group | Standard CPAP Followed by CPAP-Flex | CPAP-Flex Followed by Standard CPAP
Started | 155 | 162
Received Intervention | 144 | 146
Completed | 116 | 112
Not Completed | 39 | 50
Not completed — Physician Decision | 2 | 3
Not completed — Withdrawal by Subject | 19 | 20
Not completed — Lost to Follow-up | 18 | 27
Period: Period 2 -Cross to Alternate Arm
Arm/Group | Standard CPAP Followed by CPAP-Flex | CPAP-Flex Followed by Standard CPAP
Started | 116 | 112
Received Intervention | 103 | 95
Completed | 99 | 89
Not Completed | 17 | 23
Not completed — Lost to Follow-up | 13 | 17
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: Participants assigned to the treatment arm.
Groups:
- All Study Participants: Participants who were randomized to receive either standard CPAP or CPAP-Flex.
Arm/Group | All Study Participants
Number analyzed (Participants) | 317
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 288
  >=65 years | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.29 (8.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 282
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45
  Not Hispanic or Latino | 264
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 32
  White | 227
  More than one race | 33
  Unknown or Not Reported | 13
Apnea and Hypopnea Index (AHI4%) [Mean (Standard Deviation); unit: Events/hour] — Apneas were scored when there was a reduction in airflow to less than 10% of baseline. Hypopneas4% were scored for >30% reduction in airflow associated with 4% or more decrease in oxygen saturation. AHI4% was calculated as apneas+hypopneas4% divided by total valid recording time.
  Events/hour | 17.01 (14.42)
Total Nasal Resistance [Count of Participants; unit: Participants] — Awake nasal resistance was measured using 4-phase-rhinomanometery (RhinoLab GmbH, Rendsburg, Germany) Total nasal resistance was calculated 1/[1/Rleft + 1/Rright] and then log transformed. Total nasal resistance (TNR) measured supine was used to stratify resistance using the median value of log[TNR]=0.8. Population: TNR measurement was missing for 16 subjects at baseline.
  Participants
    number analyzed (Participants) | 301
    High Nasal Resistance (LogTNR>0.8) | 132
    Low Nasal Resistance (LogTNR<=0.8) | 169

OUTCOME MEASURES:

1. Primary Outcome: Adherence to CPAP Pre-crossover
Description: The use (number of hours per night) will be compared between standard CPAP and CPAP flex. Results are based on the first treatment period only (pre-crossover).
Time Frame: 5 weeks after initiation of treatment
Population: Subjects who received the allocated treatment (i.e., turned on the PAP device). The difference between the number allocated and the number of analyzed is the result of some subjects (n=11 in CPAP and n=16 in C-Flex) who did not turn on the device despite taking it home. These were assumed to have NOT received the allocated treatment.
Measure: Median (Inter-Quartile Range); unit: Hours/night
Groups:
- CPAP-Flex: Use of CPAP-Flex (continuous positive airway pressure) device with decreased pressure during expiration for 4 weeks to improve breathing during sleep
  CPAP - Flex: Use of Philips Respironics REMstar Auto A-Flex in C-Flex mode
Arm/Group | Standard CPAP | CPAP-Flex
Number analyzed (Participants) | 144 | 146
Hours/night | 1 [0 to 3.32] | 0.89 [0 to 3.17]

2. Primary Outcome: Adherence to CPAP Overall Study
Description: The use (number of hours per night) will be compared between standard CPAP and CPAP flex. Results are based on both periods.
Time Frame: 9 weeks after initiation of treatment
Population: Subjects who received the allocated treatment (i.e., turned on the PAP device) in either the first treatment period or the second treatment period.
Measure: Median (Inter-Quartile Range); unit: Hours/night
Arm/Group | Standard CPAP | CPAP-Flex
Number analyzed (Participants) | 239 | 249
Hours/night | 1.03 [0 to 3.33] | 0.8 [0 to 2.86]

3. Secondary Outcome: CPAP Efficacy
Description: Efficacy will be evaluated by measuring the residual apnea and hypopnea index (AHI) while on treatment. The efficacy of standard CPAP and CPAP-flex will be compared. Results are based on the first treatment period only (pre-crossover).
Time Frame: 5 weeks after initiation of treatment
Population: Subjects who received treatment (turned on the PAP device). An additional 48 subjects on CPAP and 53 on CPAP-FLex were not analyzed as an AHI could not be generated during the analysis period due to insufficient use.
Measure: Mean (Standard Deviation); unit: Events/hour
Arm/Group | Standard CPAP | CPAP - Flex
Number analyzed (Participants) | 96 | 93
Events/hour | 2.89 (3.06) | 3.12 (2.95)

4. Secondary Outcome: CPAP Efficacy
Description: Efficacy will be evaluated by measuring the residual apnea and hypopnea index (AHI) while on treatment. The efficacy of standard CPAP and CPAP-flex will be compared. Results are based on both treatment periods.
Time Frame: 9 weeks after initiation of treatment
Population: Subjects who received the allocated treatment (i.e., turned on the PAP device; N=239 for CPAP and N=249 for CPAP Flex). An additional 82 subjects on CPAP and 102 subjects on CPAP-Flex were not analyzed as an AHI could not be generated during the analysis period due to insufficient use.
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Standard CPAP | CPAP-Flex
Number analyzed (Participants) | 157 | 147
events/hour | 2.71 (2.76) | 2.94 (2.65)

5. Other Pre Specified Outcome: Adherence to CPAP Overall Study, Subjects With High Nasal Resistance
Description: The use (number of hours per night) will be compared between standard CPAP and CPAP flex for subjects with high total nasal resistance (logTNR>0.8). The analysis is based on both periods.
Time Frame: 9 weeks after initiation of treatment
Population: Subjects with high total nasal resistance who received the allocated treatment (i.e., turned on the PAP device) in either the first treatment period or in the second treatment period.Total nasal resistance data are missing for 8 subjects.
Measure: Mean (95% Confidence Interval); unit: Hours/night
Groups:
- Standard CPAP: Participants were first treated with standard CPAP (continuous positive airway pressure with constant pressure) using a REMstar Auto A-flex in standard CPAP therapy either in the first treatment period or in the second treatment period.
- CPAP-Flex: Participants were treated with CPAP-Flex (continuous positive airway pressure with a decrease in pressure during expiration) using a REMstar Auto A-flex in C-Flex either in the first treatment period or in the second treatment period.
Arm/Group | Standard CPAP | CPAP-Flex
Number analyzed (Participants) | 105 | 110
Hours/night | 2.08 [1.60 to 2.55] | 1.75 [1.31 to 2.20]

6. Other Pre Specified Outcome: Adherence to CPAP Overall Study, Subjects With Low Nasal Resistance
Description: The use (number of hours per night) will be compared between standard CPAP and CPAP flex for subjects with low total nasal resistance (logTNR<=0.8). The analysis is based on both periods.
Time Frame: 9 weeks after initiation of treatment
Population: Subjects with low total nasal resistance who received the allocated treatment (i.e., turned on the PAP device) in either the first treatment period or in the second treatment period. Total nasal resistance data are missing for 8 subjects.
Measure: Mean (95% Confidence Interval); unit: Hours/night
Groups:
- Standard CPAP: Participants were treated with standard CPAP (continuous positive airway pressure with constant pressure) using a REMstar Auto A-flex in standard CPAP therapy either in the first treatment period or in the second treatment period.
- CPAP - Flex: Participants were treated with CPAP-Flex (continuous airway pressure with a decrease in pressure during expiration) using a REMstar Auto A-flex in C-Flex either in the first treatment period or in the second treatment period.
Arm/Group | Standard CPAP | CPAP - Flex
Number analyzed (Participants) | 126 | 131
Hours/night | 1.81 [1.44 to 2.18] | 1.55 [1.22 to 1.88]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 2 months after the start of the trial.
Arm/Group | Standard CPAP | CPAP - Flex
All-Cause Mortality (participants affected / at risk) | 0/267 | 0/278
Serious Adverse Events (participants affected / at risk) | 0/267 | 0/278
Other Adverse Events (participants affected / at risk) | 0/267 | 0/278

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2016-05-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT01753999/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/99/NCT01753999/SAP_002.pdf
  • Informed Consent Form (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT01753999/ICF_003.pdf